CLINICAL TRIAL: NCT07090031
Title: Perioperative Treatment With TAS-102 in Combination With Oxaliplatin for Locally Advanced Rectal Cancer: A Single-arm, One Center Study
Brief Title: Perioperative Treatment With TAS-102 in Combination With Oxaliplatin for Locally Advanced Rectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Principal Investigator, Youxin Ji, director, Qingdao Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY202502802
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: EFS; pCR Rate
Keywords: TAS-102; Oxaliplatin; local advanced rectal cancer; concurrent chemoradiotherapy
MeSH Terms: interventions — trifluridine tipiracil drug combination; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAS-102 in combination with oxaliplatin and concurrent radiotherapy (Experimental)
  Interventions: Drug: TAS-102 in combination with oxaliplatin

INTERVENTIONS:
Drug: TAS-102 in combination with oxaliplatin — Induction : TAS102 35mg/m2, twice a day for 5 days, on 1st, 3rd, 5th week; Oxliplatin 85mg/m2 on 1st and 2nd week; Rectal radiotherapy 50GY/25f in 5 weeks. 2 weeks no treatment.
  Consolidation: TAS102 35mg/m2, twice a day for 5 days, every 2 weeks, Oxliplatin 85 mg/m2, every 2 weeks a cycle, for total 3 cycles. 4 weeks no treatment.
  Surgery Adjuvant chemotherapy: TAS102 35mg/m2, twice a day for 5 days, every 2 weeks, Oxliplatin 85 mg/m2, every 2 weeks a cycle, for total 16 cycles.

SUMMARY:
5-Fluorouracil (5-FU) based chemoradiotherapy is regarded a standard perioperative treatment in locally advanced rectal cancer, but the effective rate still low. We investigate oral TAS-102 plus oxaliplatin concurrent radiotherapy for stage II or III local advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are 18 years or older and have histologically confirmed adenocarcinoma of the rectum (defined as the distal border of the tumour less than 16 cm from the anal verge measured by rigid rectoscopy) with no evidence of distant metastases (identified by abdominal ultrasound or CT scan and chest radiography).

  * Patients in the adjuvant cohort have undergone R0-resection by total mesorectal excision (TME) of a pT3-4 N any or T any N positive non-metastatic rectal cancer.
  * Patients treated in the neoadjuvant cohort need to have a clinical T3-4 N any or T any N positive tumour staged by endoscopic ultrasound, provided the lower border of the tumour is located 0 - 16 cm from the anal verge measured by rigid rectoscopy and the primary tumour is deemed resectable by TME surgery on the basis of clinical assessment. Other eligibility criteria comprise: WHO status of zero or one; adequate liver, renal, and bone marrow function defined as follows: leucocyte count > 3,500/µl, thrombocyte count > 100,000/µl, hemoglobin > 10.0 g/dl; serum bilirubin < 2.0 mg/dl, serum creatinine < 2.0 mg/dl.

Exclusion Criteria:

* Prior treatment for rectal cancer, prior chemo- or immunotherapy, prior pelvic radiotherapy, or a history of other malignant diseases within the past five years with the exception of successfully treated basal carcinoma of the skin or carcinoma in situ of the uterine cervix.
* Participation in another trial, pregnancy, breast-feeding, unwillingness to use effective contraception, or a medical condition or concomitant illness which could potentially interfere with compliance to the protocol are regarded as exclusion criteria, as well.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
pCR | 24 monthss
  pathalogical complete response rate
pathologiccal complete response rate | 24 months
  tumor cell complete disappear pathologiccally

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao Central Hospital, Qingdao, China

IPD SHARING:
Plan to Share IPD: No